CLINICAL TRIAL: NCT06173726
Title: Investigator-initiated Phase I Exploratory Clinical Study of the Safety, Tolerability, and Efficacy of BST02 Injection in the Treatment of Locally Advanced/Metastatic Liver Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: BioSyngen Pte Ltd (Industry)
Collaborators: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOSG-BST02-00
Record Dates: First submitted 2023-11-29; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Locally Advanced/Metastatic Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BST02 Injection (Experimental)
  Interventions: Biological: BST02 Injection

INTERVENTIONS:
Biological: BST02 Injection — The TIL used for tumor tissue surgical sampling of qualified subjects was used to prepare BST02 injection, and the subjects who successfully received the surgical sampling were considered to be enrolled.
  In the study process, cell transfusions were recorded as day 0 of the study. On the 3rd day (D-3) before infusion of BST02 injection, it is necessary to receive eluvial pretreatment. Considering that this product is unmodified autologous T lymphocytes, previous studies have shown that low-intensity cyclophosphamide can stimulate their proliferation in vivo. Therefore, the cyclophosphamide (Cy) single-drug regimen is recommended: Cy 250mg~1.5g/m2, a single intravenous infusion

SUMMARY:
This is an open, single-arm, investigator-initiated Phase I clinical trial to evaluate the safety, tolerability, and initial efficacy of BST02 injection in patients with locally advanced / metastatic liver cancer. This study includes a dose escalation study and a dose extension study, which will observe the effects of different IL-2 injection doses on the safety and efficacy of BST02.

After signing the informed consent, the subjects will roughly go through two periods: the main study period and the long-term follow-up period. The main study period includes screening period, treatment and safety observation period, and follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including the critical value).
2. Patients with histologically or cytologically confirmed locally advanced / metastatic liver cancer (including hepatocellular carcinoma, intrahepatic bile duct carcinoma, and metastatic liver cancer). Hepatocellular carcinoma (HCC) and cholangiocarcinoma (BCLC) are either stage C or stage B that is not suitable for local treatment/local treatment progression according to Barcelona Clinic Liver Cancer (BCLC). Metastatic liver cancer is not suitable for radical surgical treatment according to the TNM stage of the primary cancer.
3. For locally advanced liver cancer, guidelines should recommend at least first-line systemic therapy (atrilizumab + bevacizumab, sindilizumab + bevacizumab analogues; Donafenib, Renvastinib, sorafenib; FOLFOX4) after failure (disease progression or intolerance), or as determined by the investigator to be unsuitable, or the patient refused to receive the standard treatment recommended by the guidelines. For metastatic liver cancer, failure (disease progression or intolerance) of at least second-line treatment recommended by guidelines, or inappropriate treatment determined by the investigator, or refusal of standard treatment is required.
4. At least one operation without radiation or other local treatment within 28 days to remove the tumor lesion with an estimated lesion volume of at least 8 cm^3, excluding necrotic areas, for the preparation of BST02 cells.
5. There is at least one measurable lesion after sampling that meets the definition of RECIST 1.1 standard, and the intrahepatic target lesion requires arterial phase enhanced imaging.
6. The Eastern Cooperative Oncology Group (ECOG) score ≤1 score.
7. Child-Pugh score of cirrhosis ≤7 points.
8. Expected survival time ≥3 months.
9. Adequate organ and bone marrow function in the assessment conducted during the screening period (within 14 days prior to TIL sampling), as defined below:

   * Blood routine: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L, Blood Platelet count (PLT) ≥90×10^9/L, Hemoglobin (Hemoglobin, ANC) ≥1.5×10^9/L HGB) ≥80 g/L (no blood transfusion or erythropoietin treatment within 14 days).
   * Liver function: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) levels ≤5× upper limit of normal value (ULN), Serum Total Bilirubin (TBil) ≤1.5×ULN, if diagnosed with Gilbert syndrome: TBil≤3×ULN.
   * Coagulation function: Activated partial thromboplastin time (APTT) ≤1.5×ULN, while International Normalized Ratio, INR), Prothrombin Time (PT) ≤1.5×ULN.
   * Renal function: Serum Creatinine (Cr) ≤1.5×ULN or Creatinine Clearance (Ccr) ≥60 mL/min (Cockcroft-Gault formula).
   * Cardiac function examination: Left ventricular Ejection Fraction (LVEF) ≥50% by echocardiography; No arrhythmias requiring treatment, Fridericia QT correction formulas (QTcF) ≤470 ms (QTcF is calculated using Fridericia's formula, That is, QTcF = QT/ (RR^0.33), RR is the standardized heart rate value, RR=60/ heart rate; If the first check is abnormal, the interval of at least 5 minutes, retest twice, take the comprehensive result/average value to judge the conformity);
   * Lung function: FEV1 percentage of predicted value (FEV1%) ≥60%.
10. Prior to tumor sampling, the adverse reactions caused by previous treatment had returned to the Common Adverse Event Evaluation Criteria (CTCAE) 5.0≤1 (except for alopecia, peripheral neurotoxicity of grade 2 or below, and other toxicities that the investigators judged to have no safety risk).
11. Consent to take effective contraceptive measures within 6 months from the signing of informed consent to TIL cell transfusion (subjects must use non-drug contraceptive measures).
12. Those who fully understand the test and voluntarily sign the informed consent and can comply with the visit and related procedures stipulated in the program.

    -

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects with a history of severe allergy to the experimental drugs including but not limited to cyclophosphamide, fludarabine, IL-2, and TIL injection components.
3. Patients with past or current hepatic encephalopathy, known to have other central nervous system metastases not effectively controlled by treatment or untreated, except those who have been treated and whose symptoms are stable, and who discontinue glucocorticoid and anticonvulsant therapy ≥4 weeks prior to preconditioning.
4. There is currently clinically significant ascites, which are defined as ascites with positive signs of ascites in physical examination or requiring intervention treatment (only those who show ascites on imaging without intervention can be included).
5. The proportion of liver occupied by tumor ≥50%, or ICG-R15≥30%.
6. Organ transplantation, hematopoietic stem cell transplantation history;
7. Other serious medical conditions that may limit participants' participation in the study, including but not limited to:

   * Poorly controlled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg after medication).
   * Poorly controlled diabetes: Fasting blood glucose levels remained above 11.1mmol/L after standard insulin treatment.
   * Unstable cardiovascular and cerebrovascular diseases: uncontrolled congestive heart failure, myocardial infarction or unstable arrhythmia or unstable angina within the last 6 months, percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; Cerebrovascular accident, transient ischemic attack, cerebral embolism, deep vein thrombosis, etc.
   * Poorly controlled respiratory diseases: pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease, etc.
   * Active autoimmune diseases requiring systemic treatment during the study: Subjects with eczema, vitiligo, psoriasis, alopecia, or Grave's disease that will not require systemic treatment within the next 2 years, other autoimmune diseases that are not expected to recur, and type 1 diabetes requiring insulin replacement therapy only were enrolled.
   * Have an active infection or active tuberculosis infection that requires systemic treatment.
   * Mental illness, other than mild depression.
8. HIV positive, or treponema pallidum antibody positive; Patients with active hepatitis B or C; Active hepatitis B is defined as hepatitis B core antibody (HBcAb) or Hepatitis B surface antigen (HBsAg) positive with HBV-DNA < 2000 IU/ml. HBsAg positive patients must receive antiviral treatment according to the "Chronic Hepatitis B Prevention and Treatment Guidelines 2019"; Active hepatitis C was defined as HCV RNA higher than the lower limit of detection.
9. Use of any immunosuppressive drugs, such as corticosteroids, in the 4 weeks prior to the tumor tissue sampling, or the presence of co-existing diseases that the investigator determined required the use of immunosuppressive drugs during the trial. However, the use of physiological doses of corticosteroids (i.e., no more than 15mg/ day of prednisone or equivalent doses of other corticosteroids) is permitted, and the use of corticosteroids for inhalation, intranasal, topical or prophylactic use of contrast media allergies is permitted.
10. Anti-tumor therapy was received before pretreatment, including anti-PD-1 / PD-L1 monoclonal antibodies, targeted drugs, chemotherapy, surgery, etc., and the last administration/treatment distance from pretreatment was less than 2 weeks. Or the above treatment-related adverse events, CTCAE classification does not return to grade 1 or stable.
11. Those who have received live vaccine within 3 months prior to screening or plan to receive live vaccine during the trial.
12. Those who had undergone major surgery within 4 weeks prior to screening or required elective surgery during the trial period (except TIL sampling).
13. Patients who had surgical complications or delayed wound healing prior to pretreatment and were judged by the investigators to be at increased risk of eluviation, TIL therapy, IL-2 adjuvant therapy, or infection.
14. diagnosed with other primary malignancies within 5 years prior to screening, excluding radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radical resection of carcinoma in situ.
15. Known alcohol, drug, or substance abuse, and other subjects deemed unsuitable for participation in the study.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-12-05 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Adverse events in D(0) to D(28) after BST02 cell reinfusion
  Occurrence and incidence
Severe Adverse Event | Serious adverse events in D(0) to D(28) after BST02 cell reinfusion
  Occurrence and incidence
Dose-Limiting Toxicity | Cell transfusion began until 28 days after cell transfusion
  Dose-Limiting Toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No